CLINICAL TRIAL: NCT06691256
Title: Preventing Medication Mismanagement in People Living with Dementia Through Automated Medication Dispensing with Facial Recognition and Video Observation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HiDO Technologies (Industry)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R44AG077737 (NIH)
Record Dates: First submitted 2024-11-10; First posted 2024-11-15 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease; Dementia; Medication Adherence; Type 2 Diabetes Mellitus (T2DM)
Keywords: people with dementia (PwD); Dementia; Alzheimer Disease; Medication Management; Medication Adherence; Type 2 diabetes mellitus
MeSH Terms: conditions — Alzheimer Disease; Dementia; Medication Adherence; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The Phase 2 study model for HiDO-ALZ uses a dual-study approach to refine and validate the platform:
  Field Efficacy Study: Building on in-clinic findings, this home-based trial enrolls participants in a 12-month randomized controlled study to assess the HiDO-ALZ's impact on medication adherence and health outcomes, such as adherence rates and biometric trends.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Field Efficacy Study - Experimental Group (Experimental): Participants in the experimental group will receive the HiDO-ALZ platform for 12 months, which provides automated medication dispensing, real-time facial recognition to ensure correct medication delivery, and biometric monitoring for blood pressure and weight. This arms plan to recruit up to 25 participants aged 65 or older, along with their caregivers, to assess the usability and human factors of the HiDO-ALZ platform.
  Interventions: Device: HiDO-ALZ
- Field Efficacy Study - Control Group (No Intervention): Participants in the control group will receive standard care without the HiDO-ALZ device. They will continue with their usual medication routines and any standard biometric monitoring methods as directed by their healthcare providers. This arms plan to recruit up to 25 participants aged 65 or older, along with their caregivers, to assess the standard of care and not using the HiDO-ALZ device.

INTERVENTIONS:
Device: HiDO-ALZ — HiDO-ALZ platform, an AI-driven medication dispensing and observation system designed to improve adherence in individuals with dementia and diabetes.
  Arms: Field Efficacy Study - Experimental Group

SUMMARY:
Globally, >47M individuals live with dementia, with new incidence of 7.7M annually. Medication mismanagement is one of the most common and concerning risk factors in people with dementia (PwD), as it leads to undertreatment, emergency room visits, hospital admissions/readmissions, and serious adverse events. 3M older U.S. adults are admitted to nursing homes due to drug-related adherence problems with costs >$14B/year. Furthermore, 30% of hospital admissions of older adults are drug related with 11% attributed to medication non-adherence and 17% to adverse drug reactions. While Alzheimer's disease (AD) & type 2 diabetes mellitus (DM) individually have considerable morbidity & mortality, they often occur together, worsening adverse outcomes, quality of life, & care costs. This is especially true as the AD/DM combination creates a complex balancing act of med management & symptom monitoring in older populations. While the goal is to keep older adults with dementia at home as long as possible, these challenges lead to untold personal & family suffering, as well as billions in potentially avoidable healthcare costs annually. The HiDO-ALZ platform will solve these challenges by automating medication administration for PwD to eliminate mismanagement, decrease caregiver burden, reduce healthcare utilization, and facilitate PwD to age in place. HiDO is being developed as an automated, AI driven medication dispensing and direct observation platform to optimize adherence. The device integrates medication dispensing, dose administration time, medication synchronization, & pair of front-facing cameras to validate the right meds, right route, right time, right dosage to the right patient (5R's). Cameras record every dose using facial recognition & provide real -time medication consumption recordings. Through cloud connectivity, providers & caregivers have access to video observation logs, dose administration time, adherence trends, & longitudinal adherence via web dashboard. Patients & caregivers can easily setup complex medication protocols in minutes using a smartphone app. The device then alerts patients and dispenses up to 7 different types of meds simultaneously, with up to 90 days of medication. Connected data sources including remote blood pressure and weight measurements, as well as electronic health record lab results and videoconferencing integrate in a single dashboard. The project will build on successful Phase I, in which the medication dispensing unit was updated with modifications for dementia, passed all bench testing, and was successfully validated in pilot usability with dementia subjects. Phase II will expand the foundation with four Aims: 1) Enhance device with remote sensors for diabetes management, expanded data integration, and video conferencing, 2) Test enhanced platform for usability in dementia subjects, 3) Transition the design to formal manufacturing process to ensure system meets performance standards and regulatory requirements & produce pre-production devices for testing, & 4) Conduct in-home clinical trial to demonstrate adherence and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 65 or older.
* Diagnosed with both dementia and diabetes, with documented difficulty in maintaining at least one health marker (such as glucose, HbA1c, cholesterol, blood pressure, or weight) within target levels over the past 18-24 months.
* Mild cognitive impairment or early-stage dementia, as verified by a Montreal Cognitive Assessment (MoCA) score between 18 and 24.

Exclusion Criteria:

* Cognitive deficits or serious mental health or medical conditions that would compromise safety or the reliability of feedback.
* Contraindications to taking low-dose Vitamin C (100 mg).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence: Percentage of Doses Taken as Prescribed Over 12 Months | Measurements are collected daily and weekly over 12 months.
  The primary outcome focuses on improving medication adherence among participants using the HiDO-ALZ system, as compared to standard care. Medication adherence is measured through the system's automated monitoring, which utilizes facial recognition to verify identity and track each dose administered. The HiDO-ALZ platform records the timing and accuracy of each dose taken, providing a comprehensive adherence rate over the study period. This adherence data will be evaluated against adherence rates in the standard care group, aiming to demonstrate the system's effectiveness in reducing missed doses and optimizing medication management for individuals with dementia.
Change in Health Biomarker: Change in Glucose Levels (mg/dL) Over 12 Months | Measurements are collected at baseline, 6 months, and 12 months for both adherence and biomarker levels.
  This outcome measures the average change in blood glucose levels for participants in the experimental group using the HiDO-ALZ system compared to the control group receiving standard care. Blood glucose levels will be measured at baseline, 6 months, and 12 months, with the change calculated as the difference from baseline to each subsequent time point.
  Unit of Measure: Milligrams per Deciliter (mg/dL)
Change in Health Biomarker: Change in HbA1c Levels (%) Over 12 Months | Measurements are collected at baseline, 6 months, and 12 months for both adherence and biomarker levels.
  This outcome measures the average change in HbA1c levels for participants in the experimental group compared to the control group. HbA1c levels will be monitored at baseline, 6 months, and 12 months, with changes calculated as the difference from baseline.
  Unit of Measure: Percentage (%)
Change in Health Biomarker: Change in Creatinine Levels (mg/dL) Over 12 Months | Measurements are collected at baseline, 6 months, and 12 months for both adherence and biomarker levels.
  This outcome measures the average change in serum creatinine levels for participants in the experimental group compared to the control group. Measurements will be taken at baseline, 6 months, and 12 months, with changes calculated from baseline values.
  Unit of Measure: Milligrams per Deciliter (mg/dL)
Change in Health Biomarker: Change in Glomerular Filtration Rate (GFR) (mL/min/1.73 m²) Over 12 Months | Measurements are collected at baseline, 6 months, and 12 months for both adherence and biomarker levels.
  This outcome measures the average change in GFR, an indicator of kidney function, for participants in the experimental group compared to the control group. Measurements will be taken at baseline, 6 months, and 12 months, with changes calculated from baseline values.
  Unit of Measure: Milliliters per Minute per 1.73 m² (mL/min/1.73 m²)

SECONDARY OUTCOMES:
Monthly Weight Tracking | Measurements are taken monthly over the 12-month study duration.
  Weight will be tracked monthly for participants in the experimental group using Bluetooth-enabled devices integrated with the HiDO-ALZ platform. The weight data, recorded in kilograms, will provide insights into any weight changes over the 12-month study period, aiding in the assessment of overall health status.
Blood Pressure Monitoring (mmHg) | Measurements are taken monthly over the 12-month study duration.
  Blood pressure will be measured monthly for each participant using Bluetooth-enabled devices connected to the HiDO-ALZ system. Data, recorded in mmHg, will include both systolic and diastolic values to monitor blood pressure trends and assess the intervention's impact on cardiovascular health over time.
Monthly Heart Rate Tracking (beats per minute) | Measurements are taken monthly over the 12-month study duration.
  Heart rate will be recorded monthly in beats per minute (bpm) for participants in the experimental group through Bluetooth-enabled devices connected to the HiDO-ALZ platform. Monthly tracking will allow for the evaluation of heart rate stability and potential changes associated with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States